CLINICAL TRIAL: NCT00402467
Title: An Oral, Direct Factor Xa Inhibitor, BAY59-7939, for Prophylaxis Against Venous Thromboembolism After Total Knee Replacement: a Dose-Ranging Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Healthcare Pharmaceutical Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10945
Record Dates: First submitted 2006-11-21; First posted 2006-11-22 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Venous Thromboembolism
Keywords: Prevention of venous thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Arm 6 (Experimental)
  Interventions: Drug: Enoxaparine
- Arm 1 (Experimental)
  Interventions: Drug: Rivaroxaban (BAY59-7939)
- Arm 2 (Experimental)
  Interventions: Drug: Rivaroxaban, (BAY59-7939)
- Arm 3 (Experimental)
  Interventions: Drug: Rivaroxaban, (BAY59-7939)
- Arm 4 (Experimental)
  Interventions: Drug: Rivaroxaban, (BAY59-7939)
- Arm 5 (Experimental)
  Interventions: Drug: Enoxaparine

INTERVENTIONS:
Drug: Rivaroxaban (BAY59-7939) — 2.5mg bid
  Arms: Arm 1
Drug: Rivaroxaban, (BAY59-7939) — 5mg bid
  Arms: Arm 2
Drug: Rivaroxaban, (BAY59-7939) — 10 mg bid
  Arms: Arm 3
Drug: Rivaroxaban, (BAY59-7939) — 20mg bid
  Arms: Arm 4
Drug: Enoxaparine — 30mg bid
  Arms: Arm 5
Drug: Enoxaparine — 30mg bid
  Arms: Arm 6

SUMMARY:
The study drug, BAY59-7939, is a new drug currently being tested in the prevention of VTE. It directly inhibits factor Xa, a blood component in the pathway which leads to coagulation (clotting of blood cells). It is available as a tablet. The purpose of this study is to compare the safety and efficacy of BAY59-7939 with the safety and efficacy of the licensed drug Enoxaparin. Enoxaparin, a so-called low molecular heparin, is approved and widely used in the area of thromboprophylaxis and will be given once daily subcutaneously. In this study 4 different doses of the investigational drug BAY59-7939 will be tested in comparison to Enoxaparin. You will receive during the study either one of the following BAY59-7939 treatments or Enoxaparin. The following doses of BAY59-7939 will be tested: Dose I ; Dose II, Dose III, Dose IV. This study will run for approximately 7 months in a number of countries. In total, up to 600 patients may participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged 18 years or above and postmenopausal female subjects
* Subjects scheduled for elective total knee replacement
* Subjects written informed consent for participation after receiving detailed written and oral information previous to any study specific procedures

Exclusion Criteria:

Related to medical history:

* Any prior DVT or PE
* Myocardial infarction (MI), TIA or ischaemic stroke within the last 6 months prior to randomization
* History of heparin-induced thrombocytopenia, allergy to heparins
* Intracerebral or intraocular bleeding within the last 6 months prior to randomization
* History of gastrointestinal disease (e.g. active peptic ulcer) with gastrointestinal bleeding within the last 6 months prior to randomization
* History or presence of gastrointestinal disease which could result in an impaired absorption of the study drug (e.g. severe active inflammatory bowel disease, short gut syndrome)
* Amputation of one leg

Related to current symptoms or findings:

* Heart insufficiency NYHA III-IV
* Congenital or acquired haemorrhagic diathesis (PT INR/aPTT not within normal limits)including patients with acquired or congenital thrombophilia

  * Thrombocytopenia (platelets < 100,000/µl)
  * Macroscopic haematuria
  * Allergy to contrast media
  * Severe hypertension (SBP > 200mmHg, DBP > 100 mmHg)
  * Impaired liver function (transaminases > 2 x ULN)
  * Impaired renal function (serum creatinine > 1.5 x ULN or decreased creatinine clearance < 30ml/min)
  * Active malignant disease
  * Presence of active peptic ulcer or gastrointestinal disease with increased risk of gastrointestinal bleeding
  * Body weight < 45 kg
  * Drug- or alcohol- abuse

Related to current treatment:

* Therapy with oral anticoagulants (e.g. phenprocoumon, warfarin-sodium, heparins and factor Xa inhibitors other than study medication) and fibrinolytic therapy
* Therapy with acetylic salicylic acid or other thrombocyte aggregation inhibitors (e.g. clopidogrel, dipyridamole and ticlopidine) should be stopped one week before enrollment. Patient not able to stop ASA therapy will be excluded
* All other drugs influencing coagulation, (exception: NSAIDs with half life < 17 hrs will be allowed)
* Systemic and topical treatment with azole compounds (e.g. ketoconazole, fluconazole, itraconazole). Azole compounds should be stopped at least four days before enrollment

Miscellaneous:

* Planned intermittent pneumatic compression during active treatment period
* Planned epidural anaesthesia with indwelling epidural catheter (spinal and epidural anaesthesia without indwelling catheter is allowed)
* Therapy with another investigational product within 30 days prior to the start of the study
* Concomitant participation in another trial or study

Removal of Subjects from Study:

A subject who withdraws is one who discontinued a clinical study for any reason.

Subjects may be withdrawn from the study for the following reasons:

* At their own request or at the request of their legally acceptable representative
* If, in the investigator's opinion, continuation in the study would be detrimental to the subject's well-being
* At the specific request of the sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 613 (Actual)
Dates: Start 2004-02; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Composite endpoints of Deep vein Thrombosis (proximal and/or distal),non fatal PE and death from all causes | 5-9 days after surgery or earlier in case of symptoms indicating deep vein Thrombosis.

SECONDARY OUTCOMES:
Incidence of DVTs (total, proximal, distal) | Day 6-10
Incidence of symptomatic VTEs | Day 6-10
The composite endpoint that results from the primary endpoint by substituting VTE related death for all deaths | Day 6-10
Incidence of symptomatic VTEs (total, PE, DVT) | Day 6-10

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (35):
- United States (14):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - La Mesa, California
  - Torrance, California
  - Aurora, Colorado
  - Jacksonville, Florida
  - Palm Beach Gardens, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Decatur, Georgia
  - Cincinnati, Ohio
  - Dallas, Texas
  - Lubbock, Texas
- Canada (21):
  - Edmonton, Alberta
  - Red Deer, Alberta
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Fredericton, New Brunswick
  - Barrie, Ontario
  - Greater Sudbury, Ontario
  - Kitchener, Ontario
  - Niagara Falls, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Peterborough, Ontario
  - Richmond Hill, Ontario
  - St. Catharines, Ontario
  - Thunder Bay, Ontario
  - Toronto, Ontario
  - Welland, Ontario
  - Charlottetown, Prince Edward Island
  - Montreal, Quebec
  - Québec, Quebec